CLINICAL TRIAL: NCT06595667
Title: Fluid Responsiveness Assessment in Adult Neurosurgical Patients Undergoing Posterior Fossa Tumor Resection in the Park Bench Position: a Comparison Between Pulse Pressure Variation (PPV) and Central Venous Pressure (CVP) Guidance
Brief Title: Fluid Responsiveness in Posterior Fossa Tumor Resection: PPV and CVP Guidance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Pathomporn Pin on, M.D., Associate Professor Pathomporn Pin on, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANE-2567-0391; Chiang Mai University (Other: Chiang Mai University)
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Posterior Fossa Tumor; Brain Tumor Adult
Keywords: Parkbench position; posterior fossa tumor; pulse pressure variation; fluid responsiveness
MeSH Terms: conditions — Infratentorial Neoplasms | interventions — Central Venous Pressure

STUDY DESIGN:
Intervention Model Description: Two study groups are parallel according to the block of four randomization.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessor received the anesthetic record form by unknown of the patient and group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulse pressure variation guidance fluid administration (Experimental): In the PPV group, fluids will be administered to maintain the PPV below 13%. If hypotension coincided with a PPV exceeding 13%, an initial bolus of 200 ml crystalloid fluid solution will be given in10 minutes. PPV reassessment occurred within the subsequent 10 minutes. Alternatively, if hypotension occurs with a PPV measuring less than 13%, vasopressors such as ephedrine at a dose of 3-6 mg or norepinephrine at a dosage of 5-10 mcg intravenously as a bolus, or norepinephrine infusion at a rate of 0.03-0.3 mcg/kg/min, will be given to sustain mean arterial pressure above 65 mmHg.
  Interventions: Procedure: Pulse pressure variation
- Central venous pressure guidance fluid administration (Experimental): In the CVP group, intraoperative fluid administration aimed to maintain CVP between 8-12 cmH2O while on mechanical ventilation, ensuring mean arterial pressure remains above 65 mmHg and heart rate within 20% of baseline.
  Interventions: Procedure: Central venous pressure

INTERVENTIONS:
Procedure: Pulse pressure variation — Fluid administration during posterior fossa surgery in the parkbench position is guided by the PPV value.
  Other Names: PPV
  Arms: Pulse pressure variation guidance fluid administration
Procedure: Central venous pressure — Fluid administration during posterior fossa surgery in the parkbench position is guided by the CVP value.
  Other Names: CVP
  Arms: Central venous pressure guidance fluid administration

SUMMARY:
To answer the question: What are the differences in intraoperative fluid administration volumes between PPV and CVP-guided strategies during posterior fossa tumor resection in the park bench position?

DETAILED DESCRIPTION:
Prospective RCT is conducted to compared the amount of fluid volume in adult patients undergoing posterior fossa surgery in park bench position.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 years and above
2. American Society of Anesthesiologists (ASA) I and II
3. Diagnosis of posterior fossa tumor requiring surgical resection in the park bench position, under general anesthesia at our hospital
4. Willing to participate in the study

Exclusion Criteria:

1. Arrhythmia
2. Significant cardiac diseases
3. Chronic obstructive airway disease
4. Elevated intra-abdominal pressure
5. Tumors prone to precipitate diabetes insipidus
6. Peripheral vascular disease
7. Pulmonary hypertension
8. Patients in sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Total intraoperative fluid administration volumes during surgery | during surgery
  fluid and blood and blood volume transfusion during surgery

SECONDARY OUTCOMES:
vital signs | during surgery, the data will be recorded every 5 minutes throughout the procedure
  blood pressure both systolic and diastolic pressure
vital signs | during the admission in neurosurgical ICU up to 3 days after surgery
  blood pressure both systolic and diastolic pressure
time to extubation | 48 hours after surgery at the neurosurgical intensive care unit
  to be able to succesfully extubated, count time period of using ventilator

OTHER OUTCOMES:
vasopressor requirement | during surgery and 48 hours at the neurosurgical ICU
  type and amount of vasoactive medication
length of neurosurgical ICU stay | from date of randomization to the day of being discharged from ICU or up to 1 week after surgery, depended on which happen first
  days of ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Pathomporn P Pin on, Associate Professor, Principal Investigator — Chiang Mai University
Locations (1):
- Chiang Mai University, Chiang Mai, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pin On P, Kacha S, Saringkarinkul A, Thanakititham N. Study protocol for a randomized controlled trial comparing pulse pressure variation (PPV) and central venous pressure (CVP) guidance for fluid responsiveness assessment in neurosurgical patients undergoing posterior fossa tumor resection in park bench position. PLoS One. 2025 Jun 2;20(6):e0324590. doi: 10.1371/journal.pone.0324590. eCollection 2025. PMID 40455866